CLINICAL TRIAL: NCT07189416
Title: The Same-Day and One -Day Laparoscopic Gastric Bypass by Use the "FundoRing" Method With Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center With Integreted Apartments: Randomased Clinical Trial
Brief Title: The Same-Day and One Day Gastric Bypass by Use the "FundoRing" Method (Same-Day_FundoRing Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Society of Bariatric and Metabolic Surgeons of Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Same-Day_FundoRing
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Outpatient Surgery; Same-Day Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Same-Day Discharge (Experimental): Laparoscopic One Anastomosis Gastric Bypass by Use the "FundoRing" method with Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center with Integrated Apartments with the Same-Day Discharge
  Interventions: Procedure: Laparoscopic One Anastomosis Gastric Bypass by Use the "FundoRing" method with Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center with Integrated Apartments
- The One -Day Discharge (Active Comparator): Laparoscopic One Anastomosis Gastric Bypass by Use the "FundoRing" method with Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center with Integrated Apartments with the One -Day Discharge
  Interventions: Procedure: Laparoscopic One Anastomosis Gastric Bypass by Use the "FundoRing" method with Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center with Integrated Apartments

INTERVENTIONS:
Procedure: Laparoscopic One Anastomosis Gastric Bypass by Use the "FundoRing" method with Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center with Integrated Apartments — Laparoscopic One Anastomosis Gastric Bypass by Use the "FundoRing" method with Enhanced Recovery Protocol and Remote Monitoring in Ambulatory Surgery Center with Integrated Apartments

SUMMARY:
Outpatient surgery means that patient have surgery and often go home the same day. Safety and utilization outcomes were similar between outpatient and inpatient bariatric surgery, and outpatient was associated with shorter hospital readmission length of stay. This outpatient type of surgery called as ambulatory surgery center (ASC), same-day surgery (SDD), or office-based surgery (OBS). Researcher hypothesize that the safety (complication) and readmision after same-day and one day discharge of outpatient use laparoscopic one anastomosis gastric bypass by the FundoRing method are similar.

The objective of this study was to assess the safety and readmision of outpatient same-day and one - night (standard) laparoscopic one anastomosis gastric bypass by use the "FundoRing" method with enhanced recovery (ERAS) protocol and remote monitoring in ambulatory surgery center (ASC) with integrated apartments.

Methods: Adult participants (n=200) are randomly allocated to one of two groups:

Experimental surgical bariatric group - the first (A) group: patients (n=100) (Same-Day_FundoRingOAGB group); Active comparator surgical bariatric group - the second (B) group: patients (n=100) (Standard_FundoRingOAGB group).

Primary Outcomes

1. Cases of "The day of discharge corresponds to the planned discharge date" or Cases without Extra length of stay (ELoS)). Extra length of stay = differences between day "the day of discharge corresponds to the planned discharge date" and day "the discharge date does not match the planned date". [Time Frame: same day discharge for first group (POD0) and one day discharge (POD1) for one day group].
2. Cases of readmission (rehospitalization) after discharge due to pain, dehydration, and other non-serios surgical complications). [Time Frame: first week].
3. Cases of transfer to an urgent care clinic [Time Frame: first week].

Secondary outcomes Change of preop and body mass index (BMI) (kg/m2) [Time Frame: preop and 12 months postop].

DETAILED DESCRIPTION:
A global shift is occurring as hospital procedures move to ambulatory surgical settings.

Nearly two-thirds of all operations are performed in outpatient facilities. Outpatient surgery means that patient have surgery and often go home the same day. Safety and utilization outcomes were similar between outpatient and inpatient bariatric surgery, and outpatient was associated with shorter hospital readmission length of stay. This outpatient type of surgery called as ambulatory surgery (AS), same-day surgery (SDD), or office-based surgery (OBS).

If the patient needs to stay in the facility overnight after surgery, some authors still consider it outpatient surgery, while others consider it as standard care with at least one-night hospitalization. Fast track bariatric (Enhanced Recovery -ERAS) surgery provaded significantly fewer co-morbidities and lower rate of complications and readmission when discharge is Early (ED) on postoperative (POD) 1 in comparison then late discharge (LD) when discharged on POD 2 or 3. Implementing enhanced recovery after surgery (ERAS) protocols has added further benefits for laparoscopic ambulatory surgery.

Unlike office-based surgery (OBS), where operations are mainly performed under local anesthesia, ambulatory surgical centers (ASCs) require specialized equipment or deeper anesthesia techniques for more complex outpatient metabolic and bariatric surgery.

Ambulatory/outpatient metabolic and bariatric surgery provides significant economic benefits by reducing overall health care costs through more effective treatment of obesity-related conditions such as 2 types diabetes, hypertension, and high cholesterol, resulting in reduced medication use and length of stay (LoS) in the surgical center. And can reduce the risk of infection and hospital-acquired complications, offer greater comfort during recovery.

Patients undergoing laparoscopic bariatric procedures can be safely discharged on the day of their procedure without increased incidence of mortality, reoperation, or readmission.

Researcher hypothesize that the safety (complication) and readmision after same-day and one-day (night) discharge outpatient use laparoscopic one anastomosis gastric bypass by the FundoRing method are similar.

The objective of this study was to assess the safety and readmision of outpatient same-day and one - day laparoscopic one anastomosis gastric bypass by use the "FundoRing" method with enhanced recovery (ERAS) protocol and remote monitoring in ambulatory surgery center (ASC) with integrated apartments .

ELIGIBILITY:
Inclusion Criteria:

* Obesity with a body mass index (BMI) from 30 to 50 kg / m2;
* Type 2 diabetes mellitus with good drug control or without the need for drug correction;
* Metabolic syndrome (MS), including insulin resistance (prediabetes), dyslipidemia, hypertriglyceridemia, with compensated arterial hypertension.
* Patients with MS should correspond to ASA condition 1-2. Only mild comorbidities without significant functional limitations. Well-controlled diabetes / hypertension, not severe lung diseases.
* Absence of severe hepatomegaly and / or low score on the rating scale for conditions for surgery.
* Absence or presence of GERD grade A or B (according to the Los Angeles classification);
* Absence or presence of a hernia of the esophageal opening up to 5 cm.
* No need for other simultaneous interventions other than hiatoplasty (cruroraphy) for GERD.

Exclusion Criteria:

* ASA condition 3-4
* Obesity with a body mass index (BMI) more 50 kg / m2
* Refusal of randomization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Cases of "The day of discharge corresponds to the planned discharge date"or Cases without Extra length of stay (ELoS)). | Same postoperative day (POD 0), 1 postoperative day (POD 1)
  Cases of the extra length of stay in Same-Day and One-Day groups after intervention
Case of readmission | first week
  Cases of rehospitalization (Readmission)
Cases of transfer to an urgent care clinic | first week
  Cases of transfer to an urgent care clinic after serious complication

SECONDARY OUTCOMES:
Change of preop and body mass index | preop and 12 months postop].
  Change of preop and body mass index (BMI) (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Oral Ospanov, Professor, Principal Investigator — The Society of Bariatric and Metabolic Surgeons of Kazakhstan
Locations (1):
- Oral Ospanov, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ospanov O, Sultanov K, Koikov V, Zharov N, Dildabekov Z, Shakenov A, Yelembayev B, Duysenov G, Ospanova S. The Same-Day_FundoRing trial: protocol for a randomized controlled clinical trial of the same-day discharges after "FundoRing" gastric bypass for obesity patients in ambulatory surgery center with integrated apartments. Trials. 2026 Feb 9. doi: 10.1186/s13063-026-09530-9. Online ahead of print. PMID 41656264